CLINICAL TRIAL: NCT04637516
Title: Evaluation of an Updated Version of the Program "BlinkBlink" for Alleviation of Dry Eye Symptoms Induced by Computer Work
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Sciences and Arts Northwestern Switzerland (Other)
Responsible Party: Principal Investigator, Daniela Nosch, Professor, University of Applied Sciences and Arts Northwestern Switzerland
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-00378
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Dry Eye Syndromes; Computer Vision Syndrome
Keywords: dry eye disease; computer work; computer vision syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Subjects use two versions of the program for a set duration, separated by a washout phase. The order of versions applied is randomised.
Who Masked: Investigator
Masking Description: The investigator does not know the order of versions tested by participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Programme Version 60 sec frequency (Active Comparator): This version of the program "BlinkBlink" has a presentation frequency of 60 sec
  Interventions: Device: Animation program "BlinkBlink"
- Programme Version 300 sec frequency (Placebo Comparator): This version of the program "BlinkBlink" has a presentation frequency of 300 sec
  Interventions: Device: Animation program "BlinkBlink"

INTERVENTIONS:
Device: Animation program "BlinkBlink" — Computer program that presents horizontal bars on the computer screen that move from above and below towards each other, mimicking a blink movement.

SUMMARY:
The program "BlinkBlink" was developed to alleviate dry eye symptoms during prolonged computer work. This study aimed to show subjective and objective improvement of dry eye problems in a sample size of office workers

DETAILED DESCRIPTION:
The increased use of digital devices and the resulting increase in near work has increased the prevalence of dry eye disease (DED).

Studies show that blink frequency reduced considerably during computer work, hence the tear film is spread less regularly over the anterior surface of the eye giving rise to an unstable tear film. This may lead to tired, dry eyes.

The aim of this study was to observe if the tear film quality and dry eye symptoms may improve with the use of the computer animation program "BlinkBlink" during prolonged computer work. Participating subjects test two versions of the program, whereby one version applies the animation in a much lower frequency, hence serving as a near placebo version. The testing order of the versions is randomized.

The variables tested in this study are non-invasive tear film break up (NIBUT) and subjective dry eye symptoms with the Ocular Surface Disease Index (OSDI) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* duration of computer work of at least six hours per day during at least four days per week
* OSDI score ≥ 18
* no active pathology on the anterior eye
* Snellen visual acuity of ≥ 0.8.

Exclusion Criteria:

* acute systemic disease
* contact lens wear
* asthenopia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2018-08-17 (Actual)

PRIMARY OUTCOMES:
Subjective improvement of dry eyes | 14 days
  subjective improvement with OSDI questionnaire
objective improvement of dry eyes | 14 days
  objective improvement of tear film quality (NIBUT)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Optometry, FHNW, Olten, Canton of Solothurn, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nosch DS, Foppa C, Toth M, Joos RE. Blink Animation Software to Improve Blinking and Dry Eye Symptoms. Optom Vis Sci. 2015 Sep;92(9):e310-5. doi: 10.1097/OPX.0000000000000654. PMID 26164310